CLINICAL TRIAL: NCT00047047
Title: A Phase I Trial Of Gemcitabine, 17-Allylaminogeldanamycin (17-AAG) And Cisplatin In Advanced Solid Tumor Patients
Brief Title: Tanespimycin, Gemcitabine Hydrochloride, and Cisplatin in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01429; MC0111; MAYO-MC0111; CDR0000257247; NCI-5291; U01CA069912 (NIH)
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Gemcitabine; tanespimycin; Cisplatin

ARMS (1):
- Treatment (tanespimycin, gemcitabine hydrochloride, cisplatin) (Experimental): Cohort A (closed to accrual as of 3/2/04)*: Patients receive escalating doses of gemcitabine hydrochloride intravenously (IV) over 30 minutes, tanespimycin IV over 1 hour, and cisplatin IV over 2 hours on days 1 and 8. NOTE: *The maximum tolerated dose (MTD) of this 3-drug combination has been determined as of 3/2/04.
  Cohort B (closed to accrual as of 3/2/05): Patients receive gemcitabine hydrochloride** IV over 30 minutes, tanespimycin IV over 1 hour, and cisplatin** IV over 2 hours on days 1 and 8.
  Cohort C: Patients receive gemcitabine hydrochloride** IV over 30 minutes and tanespimycin IV over 1-2 hours on days 2 and 9.
  Cohort D: Patients receive cisplatin** IV over 2 hours and tanespimycin IV over 1-2 hours on days 1 and 8.
  Cohort E: Patients receive gemcitabine hydrochloride***, tanespimycin***, and cisplatin*** as in cohort B.
  Continued (see detailed description)
  Interventions: Drug: gemcitabine hydrochloride; Drug: tanespimycin; Drug: cisplatin; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Drug: tanespimycin — Given IV
  Other Names: 17-AAG
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects, best way to give, and best doses of tanespimycin with or without gemcitabine hydrochloride and cisplatin in treating patients with advanced solid tumors. Drugs used in chemotherapy, such as tanespimycin, gemcitabine hydrochloride, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Using more than one drug (combination chemotherapy) may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximally tolerated dose (MTD) of 17-AAG (tanespimycin) when given on days 1 and 8 of every 3 weeks cycle in combination with Gemzar (gemcitabine hydrochloride) and CDDP (cisplatin) (cohorts A, B, and E).

II. To determine the MTD of 17-AAG plus Gemzar when Gemzar is given on days 1 and 8 and 17-AAG is given on days 2 and 9 every 3 weeks (cohort C).

III. To determine the MTD of 17-AAG plus CDDP when given on days 1 and 8 every 3 weeks (cohort D).

IV. To define the dose-limiting toxicity of 17-AAG when used in combination with Gemzar and CDDP.

V. To assess the effect of 17-AAG on surrogate markers when used in combination with Gemzar and CDDP.

VI. To report any responses observed.

OUTLINE: This is a dose-escalation study. Patients are assigned to 1 of 3 treatment cohorts.

Cohort A (closed to accrual as of 3/2/04)*: Patients receive escalating doses of gemcitabine hydrochloride intravenously (IV) over 30 minutes, tanespimycin IV over 1 hour, and cisplatin IV over 2 hours on days 1 and 8. NOTE: *The maximum tolerated dose (MTD) of this 3-drug combination has been determined as of 3/2/04.

Cohort B (closed to accrual as of 3/2/05): Patients receive gemcitabine hydrochloride** IV over 30 minutes, tanespimycin IV over 1 hour, and cisplatin** IV over 2 hours on days 1 and 8.

Cohort C: Patients receive gemcitabine hydrochloride** IV over 30 minutes and tanespimycin IV over 1-2 hours on days 2 and 9.

Cohort D: Patients receive cisplatin** IV over 2 hours and tanespimycin IV over 1-2 hours on days 1 and 8.

Cohort E: Patients receive gemcitabine hydrochloride***, tanespimycin***, and cisplatin*** as in cohort B.

In all cohorts, courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 3 months.

NOTE: **Gemcitabine hydrochloride and cisplatin dosage is constant, while 17-AAG is escalated in cohorts B, C, and D.

NOTE: ***Gemcitabine hydrochloride dosage is constant, 17-AAG is started at a higher dose level than all other cohorts, and cisplatin dosage is escalated in cohort E.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of cancer that is now considered clinically unresectable
* Absolute neutrophil count (ANC) >= 1500/uL
* Platelets (PLT) >= 100,000/uL
* Total bilirubin =< 2 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) =< 2.5 x ULN
* Creatinine =< 1.5 x ULN
* Alkaline phosphatase =< 2 x ULN or =< 5 x ULN if liver involvement
* Hemoglobin (Hgb) >= 9.0 g/dL
* Ability to provide informed consent
* Willingness to return to Mayo Clinic Rochester for follow up
* Life expectancy >= 12 weeks
* Willingness to provide all biologic specimens as required by the protocol; this is the mandatory translational research component
* Prior treatment with gemcitabine or cisplatin or both is allowed
* Patients who have had prior anthracycline must have a normal ejection fraction on multi gated acquisition scan (MUGA)
* Women of childbearing potential only: negative serum pregnancy test done =< 7 days prior to registration

Exclusion Criteria:

* Known standard therapy for the patient's disease that is potentially curative or definitely capable of extending life expectancy
* ECOG performance status (PS) 2, 3 or 4
* Uncontrolled infection
* Any of the following prior therapies:

  * Chemotherapy =< 4 weeks prior to study entry
  * Mitomycin C/nitrosoureas =< 6 weeks prior to study entry
  * Immunotherapy =< 4 weeks prior to study entry
  * Biologic therapy =< 4 weeks prior to study entry
  * Radiation therapy =< 4 weeks prior to study entry, or any radiation that potentially included the heart in the field (e.g., mantle)
  * Radiation to > 25% of bone marrow
  * Radiopharmaceuticals
  * Chest radiation
* Failure to fully recover from acute, reversible effects of prior chemotherapy regardless of interval since last treatment
* Significant cardiac disease including:

  * Heart failure that meets New York Heart Association classification III or IV
  * History of myocardial infarction =< one year of study entry
  * Uncontrolled dysrhythmias or requiring antiarrhythmic drugs, or
  * Poorly controlled angina
* Active ischemic heart disease =< 12 months prior to study entry
* Congenital long QT syndrome
* Left bundle branch block
* Central nervous system (CNS) metastases or seizure disorder
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception (condoms, diaphragm, injections, intrauterine device [IUD], or abstinence, etc.) Note: Concurrent use of oral contraceptives is contraindicated
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation)
* History of serious allergic reactions to eggs
* Concurrent use of drugs known to be inhibitors of the 3A4 enzyme
* >= grade 2 peripheral neuropathy, as defined by the National Cancer Institute (NCI) Common Toxicity Criteria (CTC) version 2.0
* Significant underlying pulmonary disease as manifested by requirement for oxygen or pulmonary fibrosis on chest x-ray
* Use of concomitant medications that prolong or may prolong corrected QT interval (QTc)
* History of serious ventricular arrhythmia (ventricular tachycardia [VT] or ventricular fibrillation [VF], >= 3 beats in a row), QTc >= 450 msec for men and 470 msec for women, or left ventricular ejection fraction (LVEF) =< 40% by MUGA
* Patients with symptomatic pulmonary disease requiring medication including the following: dyspnea, dyspnea on exertion, paroxysmal nocturnal dyspnea, oxygen requirement and significant pulmonary disease, including chronic obstructive/restrictive pulmonary disease; note: patients that meet the Medicare criteria for home oxygen should be excluded from the protocol
* Patients with a prior history of cardiac or pulmonary toxicity after receiving anthracyclines such as doxorubicin, daunorubicin, mitoxantrone, bleomycin or carmustine (BCNU)
* Patients with greater or equal to grade 2 pulmonary or cardiac symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2002-08; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
MTD of tanespimycin, gemcitabine hydrochloride, and cisplatin, determined by incidence of dose-limiting toxicity (DLT) graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | 21 days
Adverse events, graded according to NCI CTCAE version 3.0 | Up to 30 days after completion of study treatment
  The number and severity of all adverse events (overall, by dose-level, and by tumor group) will be tabulated and summarized within each cohort. The grade 3+ adverse events will also be described and summarized in a similar fashion. This will provide an indication of the level of tolerance for this treatment combination within each cohort. Overall toxicity incidence as well as toxicity profiles by dose level, patient and tumor site will be explored and summarized. Frequency distributions and other descriptive measures will form the basis of the analysis of these variables.

SECONDARY OUTCOMES:
Number of responses, determined according to modified Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 3 months after completion of study treatment
  Responses will be summarized (overall and by tumor type) by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease within each cohort.
Heat shock protein (HSP)70 and HSP90 client protein expression | Baseline, 6, and 25 hours after start of infusion on days 1 and 8 of course 1 (cohorts B & D); prior to gemcitabine hydrochloride on day 1; pre-dose, 6, and 25 hours post-tanespimycin dose on day 2 (cohort C)
  Descriptive statistics and simple scatterplots will form the basis of presentation of these data. The expression levels of these proteins will be summarized at the different time points as well as percent change in their levels compared (overall and within each patient) between the different time points to assess potential drug interaction. Correlations between these laboratory correlate values and other outcome measures like toxicity and response will be carried out in an exploratory manner.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Erlichman, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States